CLINICAL TRIAL: NCT04816851
Title: Autologous Pericardial Tricuspid Reconstruction of Aortic Valve Leaflets (Ozaki Procedure) in Aortic Valve Diseases
Brief Title: Aortic Valve Leaflets Reconstruction (Ozaki Procedure) in Aortic Valve Diseases
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Emad El-Dein Omar, specialist, Assiut University
Other Study IDs: 17200559
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ozaki group: Patients undergoing aortic valve reconstruction using autologous pericardium (OZAKI technique) at Assiut University Hospitals in conjunction with Al-Nas hospital in cairo.
  Interventions: Procedure: OZAKI technique

INTERVENTIONS:
Procedure: OZAKI technique — an alternative way of repairing aortic valve, involving the use of autologous pericardium for the aortic leaflet reconstruction. Diseased leaflets are removed carefully. The distance between each commissure is measured with invented sizing apparatus. The new leaflet of the size corresponding to the measured value is trimmed with an original template from glutaraldehyde-treated autologous pericardium. Finally, the annular margin of the pericardial leaflet was running sutured with each annulus. Commissural coaptation was secured with additional sutures. The coaptation of three new leaflets were always insured with direct vision.

SUMMARY:
Prospective Cohort Study aims at elaborating the outcomes of the Tricuspid Reconstruction of Aortic valve leaflets using autologous pericardium (Ozaki procedure) in the adult and paediatric patients. A very promising technique with the potential benefits of dodging oral anticoagulation, foreign material, and suitable for patients with small aortic annuli and in infectious endocarditis.

Performing hemodynamic evaluation, assess the clinical implementation and report preliminary results at follow up .

DETAILED DESCRIPTION:
Heart valve disease signifies a severe growing public health problem in developing countries, with aortic valve stenosis being the most common issue. Heart valve disease is commonly initiated by atherosclerotic degenerative processes, congenital anomalies, or rheumatic process. Aortic valve replacement is the gold standard in the treatment of patients with severe aortic stenosis and aortic regurgitation. Mechanical valves are favoured in younger patients (<60 years) owing to longer life-time, whereas biological valves are used for elderly patients in order to evade oral anticoagulation.

Options for aortic valve disease have improved in the last era including replacement, repair, and reconstructive options. A variety of creative techniques including leaflet extensions, neo-leaflet creation, resuspension or plication of prolapsing leaflets, and commissuroplasty to repair valves have been officially become skilled at, specially in pediatric population . In adults, the introduction of trans-catheter aortic valve inserting now permits treatment of degenerative aortic stenosis in the oldest and the highest risk patients. However, surgical treatment choices for pediatric patients with complex congenital aortic valve disease stay restricted.

In recent years, much attention has been given to the Ozaki procedure, an alternative way of repairing aortic valve, involving the use of autologous pericardium for the aortic leaflet reconstruction. Diseased leaflets are removed carefully. The distance between each commissure is measured with invented sizing apparatus. The new leaflet of the size corresponding to the measured value is trimmed with an original template from glutaraldehyde-treated autologous pericardium. Finally, the annular margin of the pericardial leaflet was running sutured with each annulus. Commissural coaptation was secured with additional sutures. The coaptation of three new leaflets were always insured with direct vision.

ELIGIBILITY:
Inclusion Criteria:

* Subject with AV disease.
* Documented symptomatic moderate or greater aortic stenosis
* small aortic annulus patients
* A symptomatic aortic insufficiency patient with left ventricular dysfunction or significant left ventricular dilatation.
* Patients with aortic regurgitation caused by: a dilated aortic annulus, conjoined cusp prolapse in bicuspid aortic valves (BAV), single cusp prolapse in tricuspid aortic valve (especially in paediatric population), and aortic valve cusp perforation from endocarditis.
* Concomitant intervention of the aortic root, Concomitant intervention of the aortic arch, Concomitant valve surgery and Concomitant intervention at congenital anomaly.

Exclusion Criteria:

* Patients with previous aortic valve surgery.
* missing informed consent
* Participation in another clinical research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing aortic valve reconstruction using autologous pericardium (OZAKI technique) at Assiut University Hospitals in conjunction with Al-Nas hospital in cairo.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
aortic transvalvular gradient | at follow up frame through one year
  analyse aortic valve stenosis or insufficiency measured by transthoracic echocardiography

SECONDARY OUTCOMES:
Duration of hospitalization | average 5-7 days
  number of days spent
number of patients developed complications | through one year
  the study will be monitored for Endocarditis, thromboembolic manifestation, intracranial hemorrhage
conduction disturbances | 6 months post operative
  the patients will be monitored for arrhythmia

OTHER OUTCOMES:
aortic valve re intervention or aortic regurge | through one year
  analyse aortic valve stenosis or insufficiency measured by transthoracic echocardiography
LV dimensions and EF%. | through one year
  Follow up Echocardiography data such as LV dimensions and EF%.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Abd Elwahab, PHD, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt